CLINICAL TRIAL: NCT00630539
Title: Efficacy and Safety of Ospemifene in the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women: A Phase II Dose Ranging, 12-Week, Randomized , Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing Oral Ospemifene 5 mg, 15 mg and 30 mg Daily Doses With Placebo
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Ospemifene in the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: Hormos Medical (Industry); QuatRx Pharmaceuticals (Industry)
Responsible Party: Shionogi Clinical Trials Administrator, Shionogi
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-50717
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-03

CONDITIONS: Atrophy; Vaginal Diseases
Keywords: Menopausal symptoms; Urogenital atrophy; Vulvar and vaginal atrophy in postmenopausal women; Vaginal atrophy
MeSH Terms: conditions — Atrophy; Vaginal Diseases | interventions — Ospemifene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Subjects on placebo (Placebo Comparator): Subjects will self-administer 1 placebo tablet daily (in the morning with food) for 12 weeks
  Interventions: Drug: Placebo
- Subjects on ospemifene 5 mg/day (Experimental): Subjects will self-administer 1 ospemifene 5 mg tablet daily (in the morning with food) for 12 weeks
  Interventions: Drug: Ospemifene 5 mg
- Subjects on ospemifene 15 mg/day (Experimental): Subjects will self-administer 1 ospemifene 15 mg tablet daily (in the morning with food) for 12 weeks
  Interventions: Drug: Ospemifene 15 mg
- Subjects on ospemifene 30 mg/day (Experimental): Subjects will self-administer 1 ospemifene 30 mg tablet daily (in the morning with food) for 12 weeks
  Interventions: Drug: Ospemifene 30 mg

INTERVENTIONS:
Drug: Placebo — 1 tablet per day, orally, in the morning, with food for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (End of therapy, Week 12).
  Arms: Subjects on placebo
Drug: Ospemifene 5 mg — 1 tablet of ospemifene 5 mg (QD), orally, in the morning, with food for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (End of therapy, Week 12).
  Arms: Subjects on ospemifene 5 mg/day
Drug: Ospemifene 15 mg — 1 tablet of ospemifene 15 mg (QD), orally, in the morning, with food for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (End of therapy, Week 12).
  Arms: Subjects on ospemifene 15 mg/day
Drug: Ospemifene 30 mg — 1 tablet of ospemifene 30 mg (QD), orally, in the morning, with food for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (End of therapy, Week 12).
  Arms: Subjects on ospemifene 30 mg/day

SUMMARY:
The purpose of the study is to assess the efficacy, safety and tolerability of Ospemifene 5 mg, 15 mg, and 30 mg in the treatment of VVA in postmenopausal women to find the minimum effective dose below the lowest dose of 30 mg tested earlier in Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically menopausal
* Vaginal pH greater than 5.0
* 5% or fewer superficial cells in maturation index of vaginal smear

Exclusion Criteria:

* Evidence of endometrial hyperplasia, cancer or other pathology
* Abnormal PAP smear
* Uterine bleeding of unknown origin or uterine polyps
* Current vaginal infection requiring medication
* Use of hormonal medications
* Clinically significant abnormal gynecological findings other than signs of vaginal atrophy

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers in Finland. First patient was enrolled on August 09, 2007 and last patient completed on February 11, 2008
Pre-assignment Details: The study population included postmenopausal women 40 to 80 years of age with a diagnosis of vulvar and vaginal atrophy (VVA) assessed by the maturation index (MI) of vaginal smear and vaginal pH at baseline
Groups:
- Subjects on Placebo: Subjects took 1 placebo tablet daily (in the morning with food) for 12 weeks
- Subjects on Ospemifene 5 mg/Day: Subjects took 1 ospemifene 5 mg tablet daily (in the morning with food) for 12 weeks
- Subjects on Ospemifene 15 mg/Day: Subjects took 1 ospemifene 15 mg tablet daily (in the morning with food) for 12 weeks
- Subjects on Ospemifene 30 mg/Day: Subjects took 1 ospemifene 30 mg tablet daily (in the morning with food) for 12 weeks
Period: Overall Study
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Started | 34 | 33 | 29 | 30
Completed | 33 | 29 | 28 | 27
Not Completed | 1 | 4 | 1 | 3
Not completed — Adverse Event | 1 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day | Total
Number analyzed (Participants) | 34 | 33 | 29 | 30 | 126
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (6.0) | 61.5 (5.6) | 63.4 (7.1) | 62.0 (6.8) | 62.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 29 | 30 | 126
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Participants | 34 | 33 | 29 | 30 | 126
Weight [Mean (Standard Deviation); unit: kg] | 69.6 (10.1) | 66.5 (10.6) | 68.7 (13.5) | 65.9 (7.4) | 67.7 (10.4)
Height [Mean (Standard Deviation); unit: m] | 1.609 (0.049) | 1.636 (.051) | 1.641 (.062) | 1.617 (.058) | 1.626 (0.055)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.89 (3.95) | 24.78 (3.44) | 25.50 (4.99) | 25.28 (3.20) | 25.61 (3.90)
Alcohol [Mean (Standard Deviation); unit: drinks/week] | 0.9 (1.9) | 1.8 (2.4) | 1.2 (1.7) | 1.5 (2.3) | 1.4 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
percentage of parabasal cells | -3.0 (30.2) | -2.8 (33.2) | -24.1 (36.7) | -26.8 (41.1)

2. Primary Outcome: Mean Change From Baseline in Percentage of Superficial Cells in Maturation Index of the Vaginal Smear
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
percentage of superficial cells | 0.2 (1.5) [-3 to 5] | 0.9 (3.1) [-4 to 11] | 5.0 (9.1) [-5 to 30] | 5.6 (10.3) [-5 to 35]

3. Primary Outcome: Mean Change From Baseline in Vaginal pH
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
pH | -0.07 (0.91) | -0.37 (0.83) | -0.95 (1.02) | -1.11 (1.06)

4. Secondary Outcome: Visual Evaluation of Vagina (by Gynecological Examination)
Time Frame: Screening & Week 12
Population: ITT
Measure: Number; unit: percentage of subjects
Groups:
- Subjects on Placebo (Week 12): Subjects took 1 placebo tablet daily (in the morning with food) for 12 weeks
- Subjects on Ospemifene 5 mg/Day (Week 12): Subjects took 1 ospemifene 5 mg tablet daily (in the morning with food) for 12 weeks
- Subjects on Ospemifine 15 mg/Day (Week 12): Subjects took 1 ospemifene 15 mg tablet daily (in the morning with food) for 12 weeks
- Subjects on Ospemifene 30 mg/Day (Week 12): Subjects took 1 ospemifene 30 mg tablet daily (in the morning with food) for 12 weeks
Arm/Group | Subjects on Placebo | Subjects on Placebo (Week 12) | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 5 mg/Day (Week 12) | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifine 15 mg/Day (Week 12) | Subjects on Ospemifene 30 mg/Day | Subjects on Ospemifene 30 mg/Day (Week 12)
Number analyzed (Participants) | 34 | 34 | 33 | 33 | 29 | 29 | 30 | 30
percentage of subjects
  Petechiae-None | 14.7 | 35.3 | 24.2 | 36.4 | 10.3 | 55.2 | 10.0 | 60.0
  Petechiae-Mild | 47.1 | 29.4 | 42.4 | 39.4 | 55.2 | 24.1 | 53.3 | 30.0
  Petechiae-Moderate | 26.5 | 26.5 | 12.1 | 6.1 | 31.0 | 17.2 | 26.7 | 3.3
  Petechiae-Severe | 11.8 | 8.8 | 21.2 | 15.2 | 3.4 | 0.0 | 10.0 | 3.3
  Petechiae-Not done | 0.0 | 0.0 | 0.0 | 3.0 | 0.0 | 3.4 | 0.0 | 0.0
  Pallor-None | 8.8 | 14.7 | 6.1 | 15.2 | 13.8 | 37.9 | 6.7 | 46.7
  Pallor-Mild | 44.1 | 47.1 | 30.3 | 48.5 | 48.3 | 48.3 | 40.0 | 43.3
  Pallor-Moderate | 41.2 | 35.3 | 57.6 | 30.3 | 31.0 | 10.3 | 43.3 | 6.7
  Pallor-Severe | 5.9 | 2.9 | 6.1 | 3.0 | 6.9 | 0.0 | 10.0 | 0.0
  Pallor-Not done | 0.0 | 0.0 | 0.0 | 3.0 | 0.0 | 3.4 | 0.0 | 0.0
  Friability-None | 8.8 | 20.6 | 15.2 | 30.3 | 10.3 | 44.8 | 16.7 | 60.0
  Friability-Mild | 41.2 | 32.4 | 27.3 | 30.3 | 34.5 | 44.8 | 40.0 | 33.3
  Friability-Moderate | 38.2 | 41.2 | 36.4 | 33.3 | 48.3 | 6.9 | 23.3 | 3.3
  Friability-Severe | 11.8 | 5.9 | 21.2 | 3.0 | 6.9 | 0.0 | 20.0 | 0.0
  Friability-Not done | 0.0 | 0.0 | 0.0 | 3.0 | 0.0 | 3.4 | 0.0 | 0.0
  Vaginal dryness in the mucosa-None | 8.8 | 23.5 | 6.1 | 27.3 | 10.3 | 51.7 | 10.0 | 73.3
  Vaginal dryness in the mucosa-Mild | 47.1 | 41.2 | 21.2 | 36.4 | 41.4 | 37.9 | 43.3 | 16.7
  Vaginal dryness in the mucosa-Moderate | 38.2 | 32.4 | 63.6 | 30.3 | 37.9 | 6.9 | 33.3 | 6.7
  Vaginal dryness in the mucosa-Severe | 5.9 | 2.9 | 9.1 | 3.0 | 10.3 | 0.0 | 13.3 | 0.0
  Vaginal dryness in the mucosa-Not done | 0.0 | 0.0 | 0.0 | 3.0 | 0.0 | 3.4 | 0.0 | 0.0
  Vaginal redness in the mucosa-None | 8.8 | 20.6 | 18.2 | 39.4 | 17.2 | 51.7 | 10.0 | 53.3
  Vaginal redness in the mucosa-Mild | 52.9 | 41.2 | 33.3 | 21.2 | 48.3 | 27.6 | 50.0 | 40.0
  Vaginal redness in the mucosa-Moderate | 26.5 | 26.5 | 33.3 | 21.2 | 31.0 | 17.2 | 23.3 | 0.0
  Vaginal redness in the mucosa-Severe | 11.8 | 11.8 | 15.2 | 15.2 | 3.4 | 0.0 | 16.7 | 3.3
  Vaginal redness in the mucosa-Not done | 0.0 | 0.0 | 0.0 | 3.0 | 0.0 | 3.4 | 0.0 | 0.0

5. Secondary Outcome: Mean Change From Baseline in Vaginal pH
Time Frame: Week 4
Population: ITT
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
pH | -0.12 (0.59) | -0.26 (0.68) | -0.53 (0.83) | -0.78 (1.00)

6. Secondary Outcome: Mean Change From Baseline in Percentage of Superficial Cells in the Maturation Index
Time Frame: Week 4
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
percentage of superficial cells | 0.6 (2.7) [-4 to 9] | 0.6 (2.9) [-4 to 11] | 2.5 (5.6) [-3 to 23] | 5.0 (10.7) [-4 to 55]

7. Secondary Outcome: Mean Change From Baseline in Estradiol Levels
Time Frame: Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
nmol/L | -0.004 (0.011) | 0.004 (0.015) | -0.010 (0.026) | -0.003 (0.008)

8. Secondary Outcome: Mean Change From Baseline in Luteinizing Hormone Levels
Time Frame: Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
U/L | -1.36 (4.71) | -2.89 (5.94) | -0.34 (9.23) | -3.78 (7.34)

9. Secondary Outcome: Mean Change From Baseline in Follicle Stimulating Hormone Levels
Time Frame: Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
U/L | -10.36 (20.41) | -7.04 (10.80) | -5.99 (23.07) | -15.32 (13.13)

10. Secondary Outcome: Mean Change From Baseline in Sex Hormone Binding Globulin Levels
Time Frame: Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
nmol/L | -2.4 (10.0) | 2.9 (12.2) | 6.3 (12.5) | 18.0 (20.2)

11. Secondary Outcome: Mean Change From Baseline in Percentage of Parabasal Cells in the Maturation Index
Time Frame: Week 4
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Number analyzed (Participants) | 34 | 33 | 29 | 30
percentage of parabasal cells | -0.6 (24.1) | -0.6 (23.8) | -19.7 (27.0) | -22.0 (42.7)

ADVERSE EVENTS:
Time Frame: Throughout the study
Arm/Group | Subjects on Placebo | Subjects on Ospemifene 5 mg/Day | Subjects on Ospemifene 15 mg/Day | Subjects on Ospemifene 30 mg/Day
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/33 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 25/34 | 7/33 | 13/29 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on Placebo (N=34) | Subjects on Ospemifene 5 mg/Day (N=33) | Subjects on Ospemifene 15 mg/Day (N=29) | Subjects on Ospemifene 30 mg/Day (N=30)
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on Placebo (N=34) | Subjects on Ospemifene 5 mg/Day (N=33) | Subjects on Ospemifene 15 mg/Day (N=29) | Subjects on Ospemifene 30 mg/Day (N=30)
Influenza (Infections and infestations) | 2 | 0 | 1 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 2
Vaginitis bacterial (Infections and infestations) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 1 | 5 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Genital discharge (Reproductive system and breast disorders) | 1 | 0 | 2 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Vulvovaginal discomfort (Reproductive system and breast disorders) | 2 | 0 | 1 | 0
Hot flush (Vascular disorders) | 2 | 3 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.